CLINICAL TRIAL: NCT04333511
Title: Brain Stimulation for Patients With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Storz Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU 14/032
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): TPS first with crossover to Sham-TPS
  Interventions: Device: TPS (NEUROLITH); Device: Sham-TPS (NEUROLITH)
- Sequence 2 (Experimental): Sham-TPS first with crossover to TPS
  Interventions: Device: TPS (NEUROLITH); Device: Sham-TPS (NEUROLITH)

INTERVENTIONS:
Device: TPS (NEUROLITH) — 6 treatments of TPS over 2 weeks
Device: Sham-TPS (NEUROLITH) — 6 treatments of Sham-TPS over 2 weeks

SUMMARY:
The aim of this crossover study is to investigate the efficacy of non-invasive brain stimulation (transcranial pulse stimulation; TPS) in adults with Parkinson Disease (PD). Participants will receive 6 sessions of TPS and Sham-TPS, respectively, in random order. Motor manifestations of PD and manual dexterity will be the primary outcome measures. Outcomes will be assessed immediately post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable PD with fine skilled and/or gross motor deficits (e.g. right arm with a clinical force level >2)
* Signed written informed consent
* Monthly pregnancy test for women in childbearing years
* Age >= 18 years

Exclusion Criteria:

* Non-compliance with the protocol
* Pregnant or breastfeeding women
* Relevant intracerebral pathology unrelated to the disease (e.g. Brain tumor)
* Hemophilia or other blood clotting disorders
* Cortisone treatment within the last 6 weeks before first treatment
* Thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Motor manifestations of Parkinson Disease | Immediately post-treatment
  Motor manifestations of Parkinson Disease will be rated by an examiner using the relevant subscale (section III) of the Unified Parkinson Disease Rating Scale (UPDRS). This scale has 14 different types of ratings, with many of these ratings done independently for the different limbs (tremor at rest, action tremor, rigidity, bradykinesia, speech, facial expression, arising from a chair, posture, gait, postural stability, body bradykinesia). Each of the ratings ranges from 0 (normal) to 4 (severe manifestation). The total score for this scale ranges from 0 to 108, the sum of scores from 27 observations (Perlmutter 2009).
Motor manifestations of Parkinson Disease | 1 month post-treatment
  Motor manifestations of Parkinson Disease will be rated by an examiner using the relevant subscale (section III) of the Unified Parkinson Disease Rating Scale (UPDRS). This scale has 14 different types of ratings, with many of these ratings done independently for the different limbs (tremor at rest, action tremor, rigidity, bradykinesia, speech, facial expression, arising from a chair, posture, gait, postural stability, body bradykinesia). Each of the ratings ranges from 0 (normal) to 4 (severe manifestation). The total score for this scale ranges from 0 to 108, the sum of scores from 27 observations (Perlmutter 2009).
Manual dexterity | Immediately post-treatment
  Deficits in fine skilled movements will be assessed by the coin rotation test (Foki et al., 2010). A coin hast to be flipped with the first 3 fingers of one hand as fast as possible for 30 seconds. The number of successful half rotations will be determined.
Manual dexterity | 1 month post-treatment
  Deficits in fine skilled movements will be assessed by the coin rotation test (Foki et al., 2010). A coin hast to be flipped with the first 3 fingers of one hand as fast as possible for 30 seconds. The number of successful half rotations will be determined.

SECONDARY OUTCOMES:
Activities of daily living (ADL) | Immediately post-treatment
  ADL will be assessed using the relevant subscale (section II) of the UPDRS. The scale consists of 13 items (speech, salivation, swallowing, handwriting, cutting food and handling utensils, dressing, hygiene, turning in bed and adjusting bedclothes, falling (unrelated to freezing), freezing when walking, walking, tremor, sensory complaints related to parkinsonism). The scoring range for each item is from 0 (normal) to 4 (severe impairment). The examiner asks the patient to describe their function separately in the ON and OFF state. The responses for each of the items are therefore scored twice. These ratings are done by the examiner based upon the responses of the patient or caregiver. The total score for subscale 2 ranges from 0 to 56 (Perlmutter 2009).
Activities of daily living (ADL) | 1 month post-treatment
  ADL will be assessed using the relevant subscale (section II) of the UPDRS. The scale consists of 13 items (speech, salivation, swallowing, handwriting, cutting food and handling utensils, dressing, hygiene, turning in bed and adjusting bedclothes, falling (unrelated to freezing), freezing when walking, walking, tremor, sensory complaints related to parkinsonism). The scoring range for each item is from 0 (normal) to 4 (severe impairment). The examiner asks the patient to describe their function separately in the ON and OFF state. The responses for each of the items are therefore scored twice. These ratings are done by the examiner based upon the responses of the patient or caregiver. The total score for subscale 2 ranges from 0 to 56 (Perlmutter 2009).
Anatomical and Functional Magnetic Resonance Imaging (3 Tesla MRI) | Immediately post-treatment
  fMRI to analyze brain activation and connectivity. Anatomical data are also used for safety evaluations: to exclude bleeding or anatomical changes of the brain
Somatosensory evoked EEG Potentials (SEPs) | Immediately post-stimulation
  In selected participants, standard EEG / EP (Electroencephalography / Evoked Potential) data will be recorded for procedural optimizations, i.e. evaluation of most promising parameter settings (energy level and pulse frequency).
Bayer Activities of Daily Living Scale (B-ADL) | Immediately post-treatment
  The B-ADL scale is used to assess deficits in the performance of everyday activities. The scale's main target group is community dwelling patients who suffer from mild cognitive impairment or mild-to-moderate dementia. It comprises 25 items. Each item is scored from 1 (no difficulties at all) to 10 (always difficulties). The global B-ADL score is the arithmetic mean of all items.
Bayer Activities of Daily Living Scale (B-ADL) | 1 month post-treatment
  The B-ADL scale is used to assess deficits in the performance of everyday activities. The scale's main target group is community dwelling patients who suffer from mild cognitive impairment or mild-to-moderate dementia. It comprises 25 items. Each item is scored from 1 (no difficulties at all) to 10 (always difficulties). The global B-ADL score is the arithmetic mean of all items.
Leisure Behavior (FZV; German: Freizeitverhalten) | Immediately post-treatment
  The leisure behavior questionnaire has 25 items covering the following activities: information / entertainment, active movement, social interactions, creative activities, church / cultural / educational activities. The frequency of each activity is rated on a Likert-Scale from 0 (never) to 6 (daily). The total score (0-6) is calculated as the average of all 25 items.
Leisure Behavior (FZV; German: Freizeitverhalten) | 1 month post-treatment
  The leisure behavior questionnaire has 25 items covering the following activities: information / entertainment, active movement, social interactions, creative activities, church / cultural / educational activities. The frequency of each activity is rated on a Likert-Scale from 0 (never) to 6 (daily). The total score (0-6) is calculated as the average of all 25 items.
Montreal Cognitive Assessment (MOCA) | Immediately post-treatment
  The MOCA is a screening instrument for assessing cognitive impairment. It is scored out of 30 (higher scores represent better cognition) and contains sections on visuospatial/executive, naming, memory, attention, language, abstraction, and orientation.
Montreal Cognitive Assessment (MOCA) | 1 month post-treatment
  The MOCA is a screening instrument for assessing cognitive impairment. It is scored out of 30 (higher scores represent better cognition) and contains sections on visuospatial/executive, naming, memory, attention, language, abstraction, and orientation.
Geriatric Depression Scale - short form (GDS-15) | Immediately post-treatment
  he Geriatric Depression Scale (GDS) is a questionnaire to assess depression in the elderly population. This scale generates self-evaluation scores concerning various aspects with relevance for the depressive disease (e.g. mood, drive, anxiety). The short form contains 15 items. The GDS-15 score ranges from 0 (normal state) to 15 (severe depression).
Geriatric Depression Scale - short form (GDS-15) | 1 month post-treatment
  he Geriatric Depression Scale (GDS) is a questionnaire to assess depression in the elderly population. This scale generates self-evaluation scores concerning various aspects with relevance for the depressive disease (e.g. mood, drive, anxiety). The short form contains 15 items. The GDS-15 score ranges from 0 (normal state) to 15 (severe depression).
Beck Depression Inventory (BDI) | Immediately post-treatment
  BDI stands for the "Beck Depression Inventory". The Beck Depression Inventory (BDI) measures the severity of depression (Beck 1961). It is a 21-item questionnaire for self-evaluation with 0-3 scores per item. The total score is the sum of all items. It ranges from 0 (normal state) to 63 (severe depression).
Beck Depression Inventory (BDI) | 1 month post-treatment
  BDI stands for the "Beck Depression Inventory". The Beck Depression Inventory (BDI) measures the severity of depression (Beck 1961). It is a 21-item questionnaire for self-evaluation with 0-3 scores per item. The total score is the sum of all items. It ranges from 0 (normal state) to 63 (severe depression).

CONTACTS AND LOCATIONS:
Overall Officials: Roland Beisteiner, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foki T, Pirker W, Klinger N, Geissler A, Rath J, Steinkellner T, Hoellinger I, Gruber S, Haubenberger D, Lehrner J, Pusswald G, Trattnig S, Auff E, Beisteiner R. FMRI correlates of apraxia in Parkinson's disease patients OFF medication. Exp Neurol. 2010 Oct;225(2):416-22. doi: 10.1016/j.expneurol.2010.07.019. Epub 2010 Jul 24. PMID 20659452
- [Background] Perlmutter JS. Assessment of Parkinson disease manifestations. Curr Protoc Neurosci. 2009 Oct;Chapter 10:Unit10.1. doi: 10.1002/0471142301.ns1001s49. PMID 19802812